CLINICAL TRIAL: NCT05621863
Title: University of California (UC), Davis Dietary Biomarkers Development Center
Brief Title: Fruit and Vegetable Biomarker Discovery
Acronym: UCD-DBDC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1788772; 2021-67017-35783 (Other Grant/Funding Number: USDA)
Record Dates: First submitted 2022-11-10; First posted 2022-11-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Biomarkers
Keywords: Metabolomics; Diet; Fruit; Vegetables; Biomarker; Urine; Blood

STUDY DESIGN:
Intervention Model Description: Aim 1: crossover, Aim 2: parallel, Aim 3: observational
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Aim 1 Group 1 (Experimental): Order of Treatments:
  Meal Challenge 1, Meal Challenge 2, Meal Challenge 3
  Interventions: Other: Aim 1 Meal Challenge 1; Other: Aim 1 Meal Challenge 2; Other: Aim 1 Meal Challenge 3
- Aim 1 Group 2 (Experimental): Order of Treatments:
  Meal Challenge 1, Meal Challenge 3, Meal Challenge 2
  Interventions: Other: Aim 1 Meal Challenge 1; Other: Aim 1 Meal Challenge 2; Other: Aim 1 Meal Challenge 3
- Aim 1 Group 3 (Experimental): Order of Treatments:
  Meal Challenge 2, Meal Challenge 3, Meal Challenge 1
  Interventions: Other: Aim 1 Meal Challenge 1; Other: Aim 1 Meal Challenge 2; Other: Aim 1 Meal Challenge 3
- Aim 1 Group 4 (Experimental): Order of Treatments:
  Meal Challenge 2, Meal Challenge 1, Meal Challenge 3
  Interventions: Other: Aim 1 Meal Challenge 1; Other: Aim 1 Meal Challenge 2; Other: Aim 1 Meal Challenge 3
- Aim 1 Group 5 (Experimental): Order of Treatments:
  Meal Challenge 3, Meal Challenge 1, Meal Challenge 2
  Interventions: Other: Aim 1 Meal Challenge 1; Other: Aim 1 Meal Challenge 2; Other: Aim 1 Meal Challenge 3
- Aim 1 Group 6 (Experimental): Order of Treatments:
  Meal Challenge 3, Meal Challenge 2, Meal Challenge 1
  Interventions: Other: Aim 1 Meal Challenge 1; Other: Aim 1 Meal Challenge 2; Other: Aim 1 Meal Challenge 3
- Aim 2 Typical American Diet (Experimental)
  Interventions: Other: Aim 2 Typical American Diet
- Aim 2 Typical American Diet Plus Test Foods (Experimental)
  Interventions: Other: Aim 2 Typical American Diet Plus Test Foods
- Aim 2 Dietary Guidelines for Americans Diet Plus Test Foods (Experimental)
  Interventions: Other: Aim 2 Dietary Guidelines for Americans Diet Plus Test Foods

INTERVENTIONS:
Other: Aim 1 Meal Challenge 1 — A meal challenge will be provided that contains 1 serving of peaches and 2 servings of strawberries as a smoothie and 2 servings of tomatoes and 1 serving of carrot as a vegetable dish.
  Arms: Aim 1 Group 1; Aim 1 Group 2; Aim 1 Group 3; Aim 1 Group 4; Aim 1 Group 5; Aim 1 Group 6
Other: Aim 1 Meal Challenge 2 — A meal challenge will be provided that contains 1 serving of banana and 2 servings of peaches as a smoothie and 1 serving of tomatoes and 2 servings of green beans as a vegetable dish.
  Arms: Aim 1 Group 1; Aim 1 Group 2; Aim 1 Group 3; Aim 1 Group 4; Aim 1 Group 5; Aim 1 Group 6
Other: Aim 1 Meal Challenge 3 — A meal challenge will be provided that contains 2 serving of bananas and 1 serving of strawberries as a smoothie and 1 serving of green beans and 2 servings of carrots as a vegetable dish.
  Arms: Aim 1 Group 1; Aim 1 Group 2; Aim 1 Group 3; Aim 1 Group 4; Aim 1 Group 5; Aim 1 Group 6
Other: Aim 2 Typical American Diet — The diet will provide sufficient calories for weight maintenance and will contain refined grains and low amounts of fruits and vegetables, representative of the typical American diet. No bananas, strawberries, peaches, green beans, carrots, or tomatoes will be provided.
  Arms: Aim 2 Typical American Diet
Other: Aim 2 Typical American Diet Plus Test Foods — This diet will provide sufficient calories for weight maintenance and will contain refined grains and low amounts of fruits and vegetables, representative of the typical American diet. Bananas, strawberries, peaches, green beans, carrots, and tomatoes will be provided in amounts less than or equal to 1 serving per day each.
  Arms: Aim 2 Typical American Diet Plus Test Foods
Other: Aim 2 Dietary Guidelines for Americans Diet Plus Test Foods — This diet will provide sufficient calories for weight maintenance and will contain whole grains and high amounts of fruits and vegetables, representative of the Dietary Guidelines for Americans. Bananas, strawberries, peaches, green beans, carrots, and tomatoes will be provided in amounts greater than or equal to 1 serving per day each.
  Arms: Aim 2 Dietary Guidelines for Americans Diet Plus Test Foods

SUMMARY:
The purpose of this research is to find a set of markers in the blood and/or urine that can be linked to consumption of specific fruits and vegetables. This will allow for better understanding of the link between diet and health-related outcomes. Furthermore, the results of this study will lead to the development of new methods to evaluate the nutritional status of individuals in both community and clinical settings. Food frequency questionnaires and diaries/recalls can be affected by intentional or unintentional misreporting, and thus can create errors in determining nutritional status. This study will lead to the development of an objective way to assess the consumption of specific fruits and vegetables by the general population.

DETAILED DESCRIPTION:
The purpose of this research is to find a set of markers in the blood and/or urine that can be linked to consumption of specific fruits and vegetables. This will allow for better understanding of the link between diet and health-related outcomes. Furthermore, the results of this study will lead to the development of new methods to evaluate the nutritional status of individuals in both community and clinical settings. Food frequency questionnaires and diaries/recalls can be affected by intentional or unintentional misreporting, and thus can create errors in determining nutritional status. This study will lead to the development of an objective way to assess the consumption of specific fruits and vegetables by the general population.

This study includes 3 aims to identify and then validate urine and plasma biomarkers associated with fruit and vegetable intake. Aim 1 will use a randomized crossover dietary intervention to determine the dose and time response of metabolites in plasma and urine associated with exposure to a mixture of MyPlate fruits and vegetables. Aim 2 will use a parallel design, controlled diet intervention to determine whether the biomarkers of fruit and vegetable intake determined in Aim 1 are predictors of consumption in the context of a defined dietary pattern. Aim 3 will be a cross-sectional validation arm that determines if the biomarkers of food intake developed in Aims 1 and 2 have predictive value reflecting recent and habitual consumption of these foods in a heterogeneous and diverse population.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) 18.5-39.9 kg/m^2
* Willingness to provide urine and have blood drawn

Exclusion Criteria:

* Pregnancy or lactation
* Allergy or aversion to foods provided in test diet
* History of gastrointestinal disorders including the following:

  1. Ulcerative colitis or Crohn's disease
  2. Celiac sprue
  3. Hereditary non-polyposis colorectal cancer (HNPCC)
  4. Familial adenomatous polyposis
  5. Pancreatic disease
  6. Liver disease
* Previous gastrointestinal resection or bariatric surgery
* Bleeding disorders that preclude blood draws
* Recent hospital admissions (past 6 months) for myocardial infarction (MI), cerebrovascular accident (CVA), or congestive heart failure (CHF)
* Cardiovascular disease (CVD) under physician guided therapy that is not medically stable
* Cancer under radiation or chemotherapy treatment that is active or within 6 months of treatment
* Weight change (± 5% in the last 3 months)
* Regular alcohol intake of > 2 drinks/day (equivalent to 720 mL of beer, 240 mL of wine, or 90 mL of spirits), and unwilling to abstain during feeding periods
* Use of tobacco and/or marijuana, hookahs, e-cigarettes, or vapes and not willing to abstain during feeding periods
* Use of illicit drugs and not willing to abstain during feeding periods
* BMI >40 kg/m^2
* Regular (daily to weekly) use of over-the-counter (OTC) weight-loss aids and unwilling or unable to stop taking these during feeding periods
* Regular (daily to weekly) use of OTC anti-inflammatories and unwilling or unable to stop taking these during feeding periods
* Unwilling to stop taking OTC dietary supplements that interfere with the test foods being studied including pills, chewables, liquids or powders for the following (may continue if vitamin supplement is prescribed by a medical doctor):

  1. Protein supplements
  2. Soy
  3. Fiber
  4. Flaxseed
  5. Fish oil (including cod liver oil)
  6. Probiotics
  7. Carotenoids
  8. Selenium
  9. Other antioxidants
  10. Other phytochemicals
  11. Glucosamine
  12. Chondroitin
* Oral or IV antibiotic use in the past 6 months (could defer participation until 6 months post-completion of course of antibiotics)
* Seated blood pressure >140/90 mmHg
* Fasting clinical lab values outside of the following ranges:

  1. Fasting Glucose: 54-125 mg/dL
  2. Urea: 6-50 mg/dL
  3. Creatinine: 0.4-1.3 mg/dL
  4. Estimated Glomerular Filtration Rate (eGFR): >60 mL/min
  5. Sodium: 133-146 mmol/L
  6. Alanine Transaminase (ALT): 5-60 U/L
  7. Aspartate Aminotransferase (AST): 5-40 U/L
  8. Alkaline Phosphatase (ALP): 20-135 U/L
  9. Total Bilirubin: 0.0-1.9 mg/dL
  10. Total Protein: 5-9.0 g/dL
  11. Albumin: 3.5-5.9 d/L
  12. Low-density Lipoprotein (LDL) Cholesterol: <160 mg/dL
  13. Triglycerides: <500
  14. White Blood Cells: 3-10.5 Kl/µL
  15. Hematocrit: 35-48 g/dL (women), 37.5-49 g/dL (men)
* Current use of the following prescription medications:

  1. Diuretics
  2. Steroids (oral): daily oral any dose within 1 month of study (except for oral contraceptive pills)
  3. Opiates: any use within 1 month of study
  4. Hypolipidemic agents that affect GI or renal function (ie. fibrates)
  5. Hypoglycemic medications other than metformin (ie. insulin, SGLT2 inhibitor, α-glucosidase inhibitor)
  6. Psychiatric medications that affect metabolism/renal function (anti-psychotics, lithium)
  7. Biologics/immune modulators (ie. rheumatoid arthritis, psoriasis, other rheumatologic/hematologic active disease)
  8. Anti-coagulants (coumadin, heparin, Eliquis, etc.)
  9. HIV/HAART medications (dyslipidemia inducing)
* Inability to freely give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in urine metabolomics profile | Aim 1: day 3, 8, 13; overnight fasted and post prandial 0-2 hours, 2-4 hours, 4-6 hours, 6-8 hours, 8-24 hours. Aim 2: day 3, 9, 10; Aim 3: day 4.
  Urine metabolites will be measured by ultra-performance liquid chromatography mass spectrometry (UPLC-MS) before and after consumption of no, low, or high doses of study fruits and vegetables. Change will be assessed by the appearance of and change in levels of dietary-derived metabolites, which are candidate dietary biomarkers.
Change in plasma metabolomics profile | Aim 1: day 3, 8, 13; overnight fasted and post prandial 1 hour, 2 hour, 3 hour, 4 hour, 5 hour, 6 hour, 7 hour, 8 hour, 24 hour. Aim 2: days 3, 9, 10. Aim 3: day 4.
  Plasma metabolites will be measured by ultra-performance liquid chromatography mass spectrometry (UPLC-MS) before and after consumption of no, low, or high doses of study fruits and vegetables. Change will be assessed by the appearance of and change in levels of dietary-derived metabolites, which are candidate dietary biomarkers.

SECONDARY OUTCOMES:
Diet adherence | Aim 1: day 3, 8, 13. Aim 2: day 3, 6, and 9.
  Intake of test and non-test meals/foods will be monitored through weigh-backs by study personnel in Aim 1 and participant self report in Aim 2 to identify deviations in intake of fruits/vegetables of interest.
Habitual consumption of fruits and vegetables | Day 1
  3-month General Nutrition Assessment Food Frequency Questionnaires (GNA FFQ) will be administered at site visit 1 for each aim.
Acute consumption of fruits and vegetables | Days 1, 2, 3.
  An Automated Self-Administered 24-Hour (ASA24) 3-day food record will be obtained over 2 weekdays and 1 weekend day during Aim 3.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn M Slupsky, PhD, Principal Investigator — University of California, Davis
Locations (1):
- USDA ARS Western Human Nutrition Research Center, Davis, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) will be sent to the Data Coordinating Center (DCC) at Duke University. The DCC will make study data available to other Consortium members, including researchers at Fred Hutchinson Cancer Center and Harvard, and their affiliates in accordance with best practices for data safety and accessibility. The data may be stored and shared for future research without additional informed consent provided all identifiable private information, such as the subject's name or other identifying information are removed. Once identifying information is removed from the data, we will no longer be able to identify and destroy data belonging to participants who wish to remove their samples from future research. The final de-identified study data and results will be made publicly available, in accordance with National Institutes of Health (NIH) data sharing policies.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be embargoed until publications are complete, at which time they will be made available to the scientific community.

REFERENCES:
- [Derived] Chakraborty H, Sun Q, Bhupathiraju SN, Schenk JM, Mishchuk DO, Bain JR, He X, Sun J, Harnly J, Simmons W, Raftery D, Liang L, Newman JW, Fiehn O, Clish CB, Lampe JW, Bennett BJ, Navarro SL, Wang Y, Zheng C, Mossavar-Rahmani Y, McCullough ML, Huang Y, Shojaie A, Zhu W, Djukovic D, Sacks F, Williams J, Steinberg FM, Adams SH, Hu FB, Neuhouser ML, Slupsky CM, Maruvada P. The Dietary Biomarkers Development Consortium: An Initiative for Discovery and Validation of Dietary Biomarkers for Precision Nutrition. Curr Dev Nutr. 2025 Apr 5;9(5):107435. doi: 10.1016/j.cdnut.2025.107435. eCollection 2025 May. PMID 40641655